CLINICAL TRIAL: NCT00155740
Title: Mesothelin as a New Tumor Marker for Ovarian Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9100201610
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2005-11-28 (Estimated); Status verified 2001-10

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer; tumor marker; mesothelin
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Ovarian cancer became a more and more important disease in recent years due to its first mortality rate of gynecologic malignancies. The incidence of ovarian cancer also increased in recent year in Taiwan. The lack of symptoms, difficulties in early diagnosis, insufficient accurate tumor markers, and lack of information about ovarian tumor biology contribute to the poor prognosis in ovarian cancer patients. The prognostic parameters for ovarian carcinomas are tumor stage, histologic subtype, degree of malignancy, and residual tumor after surgical treatment. However, these factors present an incomplete picture of the tumor biology of ovarian cancer and are frequently interrelated. Thus, the identification of new biologic factors predictive of individual disease course and prognosis would be extremely useful.

Detection of tumor markers that are released into the circulation can aid in the diagnosis and/or monitoring of therapeutic responses of patients with various tumors, including carcinomas of ovary. CA125 is the most commonly used serum marker for patients with ovarian carcinoma. Although it has proven clinically valuable in monitoring the response of patients to therapy, some ovarian carcinomas do not express CA125, and CA125 often is increased in patients with inflammatory disease. Thus, there is a need for improvement, either in the form of a more specific and/or sensitive assay or an assay that uses a different marker and can be used to complement CA125 toward the goal to improve patient survival by improving diagnosis.

Mesothelin is a 40-kDa glycosylphosphatidylinositol-linked glycoprotein. In normal tissues, the expression of mesothelin has subsequently been shown to be largely restricted to mesothelial cells, although immunoreactivity has also been reported in epithelial cells of the trachea, tonsil, fallopian tube, and kidney. Mesothelin has been shown to be over-expressed in pancreatic carcinomas, gastric carcinoma and ovarian carcinoma, and it seems that mesothelin may be utilized as a new tumor marker for ovarian carcinoma. We will evaluate that if mesothelin can be a new potential tumor marker for ovarian cancer in this proposal.

DETAILED DESCRIPTION:
Incidence of Ovarian Cancer Ovarian cancer is the first mortality rate of gynecologic malignancies (1-3) and became a more and more important disease in recent years (4-6). The incidence of ovarian cancer also increased in recent year in Taiwan (7). Ovarian cancer has the highest mortality of all gynecological cancers, with an overall 5-year survival rate of only 20-30% (1). The lack of symptoms, difficulties in early diagnosis, insufficient accurate tumor markers, and lack of information about ovarian tumor biology contribute to the poor prognosis in ovarian cancer patients (8). The prognostic parameters for ovarian carcinomas are tumor stage, histologic subtype, degree of malignancy, and residual tumor after surgical treatment (9-12). However, these factors present an incomplete picture of the tumor biology of ovarian cancer and are frequently interrelated (13). Thus, the identification of new biologic factors predictive of individual disease course and prognosis would be extremely useful. From the above-mentioned data, ovarian cancer indeed is a disease that should be respected, however, there were only few of research work focusing on it in Taiwan.

Tumor marker for ovarian cancer Detection of tumor markers that are released into the circulation can aid in the diagnosis and/or monitoring of therapeutic responses of patients with various tumors, including carcinomas of ovary (14-17), prostate (18), the gastrointestinal tract (19, 20), or breast (21). CA125 is the most commonly used serum marker for patients with ovarian carcinoma (14). Although it has proven clinically valuable in monitoring the response of patients to therapy, some ovarian carcinomas do not express CA125, and CA125 often is increased in patients with inflammatory disease. Thus, there is a need for improvement, either in the form of a more specific and/or sensitive assay or an assay that uses a different marker and can be used to complement CA125 toward the goal to improve patient survival by improving diagnosis.

New potential molecule as tumor marker for ovarian cancer Mesothelin is a 40-kDa glycosylphosphatidylinositol-linked glycoprotein. It is synthesized as a precursor of molecular mass 69 kDa, which then is proteolytically processed into an N terminal secreted form of molecular mass 30 kDa and a membrane-bound form of 40 kDa (22, 23). The 30-kDa secreted form has been termed megakaryocyte potentiating factor (23). In normal tissues, the expression of mesothelin has subsequently been shown to be largely restricted to mesothelial cells, although immunoreactivity has also been reported in epithelial cells of the trachea, tonsil, fallopian tube, and kidney (24). Mesothelin has been shown to be expressed in pancreatic carcinomas(25), gastric carcinoma (26) and ovarian carcinoma (27), and it seems that mesothelin may be utilized as a tumor marker for ovarian carcinoma.

We will evaluate the amount of mesothelin in pre- and post-treatment serum samples of patients with epithelial ovarian cancer. We will also correlate the clinicopathologic items and the prognosis of ovarian cancer patients and evaluate whether mesothelin can be a new rumor marker for ovarian cancer patients.

ELIGIBILITY:
Inclusion Criteria:

- Patients with ovarian carcinoma who undergo hysterectomy, bilateral salpingo-oophorectomy, omentectomy, and appendectomy will be enrolled and the clinical data will be obtained from our hospital. All of the patients received four to six courses of adjuvant platinum-containing chemotherapy.Histologic grading was according to International Union against Cancer criteria (28). The stage of disease was classified according to the International Federation of Gynecology and Obstetrics (FIGO, 1987). Pelvic and paraaortic lymph node samplings will be performed, if the disease will be confined to within the ovary or will be without a ruptured capsule. The histopathologic data, including histologic type and histologic grade, will be evaluated by a certified pathologist. The maximal diameter of the residual tumor after surgery will be also recorded. All patients will be followed up at 3-month intervals.

Patients with ovarian endometrioma, other benign ovarian tumors receiving surgical intervention, or healthy patients without surgical intervention will be presented as normal controls.

Exclusion Criteria:

-

Ages: 15 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 250
Dates: Start 2002-01; Study Completion 2006-12

CONTACTS AND LOCATIONS:
Overall Officials: Chi-An Chen, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan